CLINICAL TRIAL: NCT04933786
Title: Digital Health Nudging - Daily Smartphone Messages to Increase Physical Activity in Adolescents With Congenital Heart Disease
Brief Title: Digital Health Nudging in Adolescents With Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Collaborators: Technical University of Munich (Other); Stiftung KinderHerz Deutschland gGmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 265/21 S
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Congenital Heart Disease
Keywords: Physical Activity Promotion; Digital Health Nudging
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Health Nudging (Experimental): During 12-week intervention period participants receive daily text messages via WhatsApp on their smartphone to encourage them to be physically active in their daily lives.
  Interventions: Behavioral: Digital Health Nudging
- Control (No Intervention): During 12-week control period participants receive no text messages.

INTERVENTIONS:
Behavioral: Digital Health Nudging — Short daily text messages with information and motivation concerning physical activity.
  Arms: Digital Health Nudging

SUMMARY:
In adolescents with congenital heart disease physical activity level is reduced which is why promotion to a more active lifestyle with an age-appropriate and modern intervention is needed. In healthy subjects digital health nudging was shown to increase physical activity. However, in adolescents with congenital heart disease such studies have not been conducted yet. In this RCT participants receive daily, short smartphone messages with the primary purpose to increase daily physical activity, which is monitored with a "Garmin vivofit jr." wearable.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12 to 18 years inclusive
* Presence of a congenital heart defect (must be moderate or complex according to ACC criteria)
* Presence of written informed consent

Exclusion Criteria:

* Cognitive impairments that inhibit patients from understanding the tasks

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 97 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Objectively measured physical activity | 25 weeks
  Physical activity is objectively assessed with the wrist worn wearable "Garmin vivofit jr.". Daily physical activity is measured on the basis of active minutes in moderate-to-vigorous intensity.

SECONDARY OUTCOMES:
Objectively measured daily step count | 25 weeks
  Daily step count is objectively assessed with the wrist worn wearable "Garmin vivofit jr.".
Activity-related self-efficacy | Baseline, after 12 weeks, after 24 weeks
  Perceived self-efficacy in the context of physical activity is measured using the German version of the Physical Activity Self-Efficacy Scale. The scale consists of eight items, each of which is answered on a five-point Likert scale.
Health-related quality of life | Baseline, after 12 weeks, after 24 weeks
  Health-related quality of life is self-assessed via the KINDL® questionnaire. The KINDL® is a generic instrument for assessing health-related quality of life in children and adolescents. The KINDL® is a short, methodologically tested and flexible measurement instrument consisting of 24 questions on the six areas of body/physis, feelings/psychology, self-assessment, family, friends and school.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Müller, PD Dr.rer.nat, Study Director — Technical university munich, Chair of preventive perdiatrics
Locations (1):
- Department of Congenital Heart Defects and Pediatric Cardiology, German Heart Center, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Willinger L, Oberhoffer-Fritz R, Ewert P, Muller J. Digital Health Nudging to increase physical activity in pediatric patients with congenital heart disease: A randomized controlled trial. Am Heart J. 2023 Aug;262:1-9. doi: 10.1016/j.ahj.2023.04.001. Epub 2023 Apr 7. PMID 37030491